CLINICAL TRIAL: NCT02651285
Title: G-CSF Supplemented Medium for IVF Embryo Culture in Patients Undergoing IVF
Brief Title: Use of G-CSF Supplemented IVF Medium in Patients Undergoing IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Principal Investigator, Fabio Scarpellini, Clinical Director, Centre for Endocrinology and Reproductive Medicine, Italy
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CRH2016/01
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Infertility; Embryo Development; IVF
Keywords: G-CSF; BLASTOCYST; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Experimental): The embryos obtained with IVF in patients included iin this arm will be incubated after fertilization with medium supplemented with G-CSF
  Interventions: Other: G-CSF medium
- CONTROL (Placebo Comparator): The embryos obtained by women undergoing IVF included in this arm will be incubated with a standard medium for IVF, and utilized as control group.
  Interventions: Other: Control

INTERVENTIONS:
Other: G-CSF medium — incubation of IVF embryos with a specific medium containing G-CSF
  Other Names: (granulokine)
  Arms: G-CSF
Other: Control — incubation of IVF embryos with a medium without G-CSF
  Arms: CONTROL

SUMMARY:
The purpose of this study is to determine whether in Assisted Reproductive Technologies the use of culture medium supplemented with G-CSF, a growth factor working on stem cells, may improve the embryo implantation and pregnancy rate in infertile patients undergoing IVF cycles.

DETAILED DESCRIPTION:
In Assisted Reproductive Technologies the rate of pregnancy for cycle and the implantation rate remain low nevertheless the improvement in the last years. In particular also in relatively young reproductive age women nevertheless the good embryos produced and transferred pregnancy rate and implantation rate remain low. Recently, it has been showed that culture medium supplemented with G-CSF, may improve the embryo outcomes in IVF. In this trial the investigators will test the potential benefits of this culture medium on embryos of patients undergoing IVF. 180 infertile women undergoing IVF no more than 37 years old will be selected. These patients will be assigned to two arms, one experimental and one other of control by a computer generated sequence. After the oocyte retrieval and fertilization by ICSI procedure, the fertilised oocyte (2PN)will cultured with the G-CSF supplemented culture medium or in normal culture in micro drop of 30microliters under oil until the day of transfer (day five or blastocyst sage embryos). A maximum of two embryos will be transferred. The pregnancy rate, implantation rate and number of blastocyst developped will be the outcomes considered

ELIGIBILITY:
Inclusion Criteria:

* infertility
* healthy condition,
* good ovarian reserve (AMH levels more than 1microg/ml)

Exclusion Criteria:

* chromosomal defects in the couple,
* metabolic diseases (diabetes, etc),
* other genetic diseases (thalassemia, cystic fibrosis, etc.)

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 12 months
  The number of patients become pregnant after IVF where G-CSF medium is used divided for the number of patients treated
implantation rate | 12 months
  The number of embryos implanted after IVF where G-CSF medium is used divided for the number of embryos transferred

SECONDARY OUTCOMES:
number of blastocyst developped | 12 months
  The number of blastocysts obtained after IVF where G-CSF medium is used divided for the number of fertilized oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Morgia, MS, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (1):
- Cerm-Hungaria, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes